CLINICAL TRIAL: NCT02249364
Title: Interest of Hypnosis Before the Induction of Anesthesia. Study in Women Submitted to One Day Gynecological Surgical Procedures
Brief Title: Hypnosis Before the Induction of Anesthesia
Acronym: Hypnose2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013/49; 2013-A01640-45 (Other: ANSM); NCT02296827 (obsolete NCT alias)
Record Dates: First submitted 2014-09-23; First posted 2014-09-25 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Anesthesia
MeSH Terms: interventions — Hypnosis; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Standard care without hypnosis session followed by closed-loop administration of propofol for anesthesia induction
  Interventions: Procedure: Control; Drug: propofol
- Hypnosis (Experimental): Hypnosis session followed by closed-loop administration of propofol for anesthesia induction
  Interventions: Procedure: Hypnosis; Drug: propofol

INTERVENTIONS:
Procedure: Control — Routine practice
  Arms: Control
Procedure: Hypnosis — Hypnosis session before induction of anesthesia
  Arms: Hypnosis
Drug: propofol — Closed-loop administration of propofol for anesthesia induction

SUMMARY:
Hypnosis may reduce patient anxiety. The main goal of this study is to determine in what extent, hypnosis decreases propofol requirement to induce induction of general anesthesia.

Two particular aspects of this study are

* the inclusion of women undergoing one day gynecological surgical procedures
* the use of a closed-loop system which delivers propofol according to bispectral index to provide induction of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Adult female patients scheduled for a one day gynecological surgical procedures under general anesthesia

Exclusion Criteria:

* pregnancy, breast feeding woman
* allergy to propofol, soy or peanuts
* history of central nervous system disease
* psychiatric affection
* hypovolemia, high cardiovascular risk
* patients with a pace-maker

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Administered dose of propofol | one hour
  Administered dose of propofol required to obtain the induction of anesthesia (bispectral index <60 for at least 30 seconds)

SECONDARY OUTCOMES:
Target plasma concentration of propofol | one hour
  Target plasma concentration of propofol corresponding to induction of anesthesia (bispectral index <60 for at least 30 seconds)
Pain of insertion of peripheral vein catheter | one hour
  Pain is assessed by two criteria:
  * withdrawal of the arm perfused (no = 0; withdrawal = 1; violent withdrawal = 2),
  * spontaneous expression (no = 0; frown = 1; grin or verbal complaint = 2)
Pain due to injection of propofol | one hour
  Pain is assessed by two criteria:
  * withdrawal of the arm perfused (no = 0; withdrawal = 1; violent withdrawal = 2),
  * spontaneous expression (no = 0; frown = 1; grin or verbal complaint = 2)
Effect of hypnosis on bispectral index | one hour
  Effect of hypnosis on bispectral index before the induction of anesthesia
Time to loss of consciousness | one hour
  Time between the beginning of injection of propofol and the loss of eyelash reflex
Hemodynamic consequences of induction of anesthesia | one hour
  Heart rate and blood pressure are measured just before induction of anesthesia and once it is realized.
Administration of a cardio-vascular agent | one hour
  Administration of ephedrine, atropine or of an hypotensive agent
Manipulation of the airway | one hour
  Necessity of a jaw thrust maneuver or of another manipulation of the airway during the induction of anesthesia
Characteristics of the hypnotic procedure evaluated by the clinician in the group "hypnosis" | one hour
  The hypnotic procedure is assessed by three criteria:
  * receptivity of the patient (yes/no),
  * rapidity of focalization procedure (very fast, fast, medium, delayed, impossible to obtain),
  * quality of the hypnotic trance (very deep, deep, medium, superficial, not obtained).
Characteristics of the hypnotic procedure evaluated by the patient in the group "hypnosis" | six hours
  The hypnotic procedure is assessed by a question : "Did you visualize the memory we talked about before the session ? (yes, no )
Characteristics of the preanesthetic management evaluated by the patient (all the patients) | Six hours
  The preanesthetic management is assessed by one criteria:"How do you rate the quality of the preanesthetic period (from the entrance in the operating room to the induction of the general anesthesia ?" (excellent, good, average, not good)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, Study Chair — Hopital Foch
Locations (1):
- Dept of Anesthesia, Hôpital Foch, Suresnes, France

REFERENCES:
- [Background] Liu N, Chazot T, Genty A, Landais A, Restoux A, McGee K, Laloe PA, Trillat B, Barvais L, Fischler M. Titration of propofol for anesthetic induction and maintenance guided by the bispectral index: closed-loop versus manual control: a prospective, randomized, multicenter study. Anesthesiology. 2006 Apr;104(4):686-95. doi: 10.1097/00000542-200604000-00012. PMID 16571963
- [Derived] Bataille A, Guirimand A, Szekely B, Michel-Cherqui M, Dumans V, Liu N, Chazot T, Fischler M, Le Guen M. Does a hypnosis session reduce the required propofol dose during closed-loop anaesthesia induction?: A randomised controlled trial. Eur J Anaesthesiol. 2018 Sep;35(9):675-681. doi: 10.1097/EJA.0000000000000751. PMID 29210845